CLINICAL TRIAL: NCT02109809
Title: A Phase I Study: Low-Dose Total Lymphoid Irradiation in the Treatment of Refractory Chronic Graft Versus Host Disease
Brief Title: Low-Dose Total Lymphoid Irradiation in Treating Patients With Refractory Chronic Graft-versus-Host Disease After Donor Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00026878; NCI-2014-00671 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97114 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-10

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Supportive Care (TLI) (Experimental): Patients undergo LD-TLI daily for 1-2 days.
  Interventions: Radiation: total nodal irradiation; Other: laboratory biomarker analysis; Other: questionnaire administration

INTERVENTIONS:
Radiation: total nodal irradiation — Undergo TLI
  Other Names: TLI; total lymphoid irradiation
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and best dose of low-dose total lymphoid irradiation (LD-TLI) in treating patients with chronic graft-versus-host disease that has not responded to treatment with steroids. LD-TLI is a procedure in which all of the body's major lymph nodes are treated with small doses of radiation in order to reset the dysfunctional immune system. LD-TLI may work as a treatment for graft-versus-host disease caused by a bone marrow or stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of total lymphoid irradiation (TLI) in cohorts of a selected population of refractory chronic graft-versus-host disease (GvHD) patients, given to cohorts with a total cumulative doses of TLI of 100, 150, 200, 250 or 300 centigray (cGy).

SECONDARY OBJECTIVES:

I. To evaluate the efficacy (failure free survival [FFS] at 6 months) of this therapy in the study population.

II. Approximate the efficacy at different dose levels using the GvHD summary scores.

TERTIARY OBJECTIVES:

I. Determine the effect of this therapy on relevant subpopulations of immune cells in an attempt to elucidate a mechanism of action.

OUTLINE: This is a dose-escalation study.

Patients undergo LD-TLI daily for 1-2 days.

After completion of study treatment, patients are followed up on day 45, at 3 and 6 months, at 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have received a prior allogeneic hematopoietic stem cell transplant (alloHSCT) for any indication and from any donor
* Patients must have a diagnosis of cGvHD, in accordance with National Institutes of Health (NIH) guidelines; patients with "overlap syndrome" are also eligible; NOTE: Patients with recurrent, late onset and/or persistent acute GvHD (alone) are not eligible
* Patients with chronic GvHD who have been exposed to two or more lines of therapy, including at least one of which was composed of a glucocorticoid and a calcineurin inhibitor are eligible.
* Patients must have active, but not rapidly progressive, refractory cGvHD; any degree of severity (as per NIH criteria) and/or pattern of organ involvement may be considered; that said, patients with more severe and/or extensive chronic GvHD are expected to be the usual candidates for therapy
* As above, GvHD should be controlled to a degree that would potentially allow no additional requirement for systemic IST before and following TLI =< -15 and >= day (d) +45, respectively
* The ability to administer protocol doses of TLI (i.e., 100, 200 or 300 cGy) without exceeding cumulative doses of radiation must be established; for patients with prior radiotherapy exposure, this determination will be made by Dr. Greven (or her designee) using published guidelines for excessive organ exposure
* Karnofsky performance status (KPS) >= 60%
* White blood cells >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 10.0 g/dL
* Platelets >= 100,000/mcL
* NOTE: If such hematologic abnormalities are present and deemed due to the process of cGvHD, such requirements may be waived with the approval of the PI
* Patients must have non-hematologic organ function as defined below:

  * Left ventricular ejection fraction (LVEF) > 40%
  * Key pulmonary function tests (PFTs) > 40%

    * No further criteria for non-hematologic organ function are specified; however, if moderate-to-severe (major) organ function is present, such should be discussed with the PI, as various degrees of non-hematologic organ dysfunction may compromise either (or both) outcomes and toxicity evaluation
    * If there is concern regarding potential reversibility of any specific organ dysfunction, this issue should be addressed by consultation with an appropriate sub-specialist
* Ability to understand and the willingness to sign an institutional review board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients with evidence of persistent or active malignancy or uncontrolled infection at the time of study entry
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Phillips, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (TLI)
Started | 4
Completed | 1
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (TLI)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events, Scored as Per Common Toxicity Criteria Version 4.0
Description: Toxicities (grade 2 and higher) will be reported as number of occurrences.
Time Frame: At day 180
Population: Only 1 participant on study treatment and there are concerns of patient privacy.
Arm/Group | Supportive Care (TLI)
Number analyzed (Participants) | 0

2. Primary Outcome: Failure Free Survival (FFS) as Assessed by Scoring for Chronic GvHD - Specific Core Measures
Description: Estimated along with 95% confidence intervals (CI). Descriptive statistics will be calculated and presented for GvHD summary scores by dose level and visit.
Time Frame: Time from baseline to date of last follow-up or failure event, assessed at day 180
Population: Only 1 participant on study treatment and there are concerns of patient privacy.
Arm/Group | Supportive Care (TLI)
Number analyzed (Participants) | 0

3. Secondary Outcome: Immunomodulatory/Immuno-suppressive Effects
Description: T, natural killer (NK)T, regulatory T cell (Treg), B, NK, dendritic cell (DC) cell subsets, cell activation status and functional potential through cytokine and chemokine expression will be identified. Descriptive statistics (with 95% confidence intervals) will be calculated at each assessment time point.
Time Frame: Up to 1 year
Population: Only 1 participant on study treatment and there are concerns of patient privacy.
Arm/Group | Supportive Care (TLI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 1 year
Description: Only 1 participant on study treatment and there are concerns of patient privacy.
Arm/Group | Supportive Care (TLI)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes